CLINICAL TRIAL: NCT04517045
Title: The Study of Dachengqi Decoction Combined With Probiotic L92 to Improve the Prognosis of Patients With Severe Abdominal Hypertension
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chengjing Gao, Chief Physician, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-20-017
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Dachengqi Decoction; Probiotic L92
MeSH Terms: interventions — dachengqi decoction

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conventional treatment group (Sham Comparator): Control the primary disease, prevent infection, reduce gastrointestinal decompression, and actively maintain organ function.
  Interventions: Other: Conventional treatment
- Conventional treatment plus L92 group (Experimental): Conventional treatment combined with L92
  Interventions: Drug: probiotic L9; Other: Conventional treatment
- Conventional treatment plus Dachengqi decoction group (Experimental): Conventional treatment combined with Dachengqi Decoction
  Interventions: Drug: Dachengqi decoction; Other: Conventional treatment
- Conventional treatment plus Dachengqi decoction plus L92 group (Experimental): Conventional treatment combined with L92 and Dachengqi Decoction
  Interventions: Drug: Dachengqi decoction; Drug: probiotic L9; Other: Conventional treatment

INTERVENTIONS:
Drug: Dachengqi decoction — Raw rhubarb 30g, Glauber's salt 30g, Citrus aurantium 20g, Magnolia officinalis 20g. The decoction was decocted uniformly in the decoction room of Xinhua Hospital, Shanghai Jiaotong University School of Medicine, and decocted 200 mL thickly, fed via nasogastric tube/nasal intestine tube and enema, 1 dose/d, and continued treatment until the end of the trial
  Other Names: probiotic L92
  Arms: Conventional treatment plus Dachengqi decoction group; Conventional treatment plus Dachengqi decoction plus L92 group
Drug: probiotic L9 — L92 2 tablets/time, tid, oral or nasal feeding
  Arms: Conventional treatment plus Dachengqi decoction plus L92 group; Conventional treatment plus L92 group
Other: Conventional treatment — Conventional treatment

SUMMARY:
Patients with severe infections, wounds (burns), and severe pancreatitis often have abdominal hypertension (IAH), which is an important objective manifestation of acute gastrointestinal failure in severe patients. Timely diagnosis and effective intervention can improve the treatment rate of patients. In the early stage, we conducted clinical exploration and observational research on the treatment of IAH with Dachengqi Decoction and Lactobacillus in the treatment of critically ill patients including the above diseases, and achieved significant clinical effects. On this basis, it is planned to verify the protective effect of Lactobacillus acidophilus L92, Dachengqi Decoction and the combination of the two on the gastrointestinal mucosal barrier function of patients with IAH and the regulation of the intestinal flora, and analyze the intestinal mucosal barrier The relationship between intestinal flora and the prognosis of IAH patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion and exclusion criteria and critically ill patients (acute severe pancreatitis, cervical spinal cord injury) who are 60 years old or older than 18 years old, expected to be mechanically ventilated in the ICU, and hospitalized for more than 48 hours, replaced intra-abdominal pressure monitoring with bladder pressure measurement, and repeated on admission The results of the three measurements are ≥12 mmHg.

Exclusion Criteria:

* Patients who have not signed the informed consent; cannot tolerate intra-abdominal pressure monitoring; pregnant women; patients after bladder surgery; systemic diseases and recent use of related drugs; previous infections, such as history of tuberculosis or PPD positive; previous high History of blood pressure, poor blood pressure control (SBP/DBP>=140mmHg); patients with severe mental illness; long-term use of traditional Chinese medicine, probiotics, gastric mucosal protectors, proton pump inhibitors, chemotherapy or immunosuppressive drugs, etc., such as admission The drug was not discontinued within the previous month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 752 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of sepsis within 7 days | six months